CLINICAL TRIAL: NCT05768594
Title: Omics in Valvular Disease: Biomarkers of Cardiac Remodeling, Left Ventricular Function, Intensive Care Unit Outcome, and Doppler Echocardiography (OVERLOAD)
Brief Title: Omics in Valvular Disease
Acronym: OVERLOAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Liuzzo Giovanna, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 2821
Record Dates: First submitted 2023-02-22; First posted 2023-03-14 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Stenosis, Aortic
Keywords: Transcatheter Aortic Valve Replacement; Surgical Aortic Valve Replacement
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Years
Biospecimen Retention: Samples With DNA — Blood Sample and Cardiology visit
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with aortic stenosis, surgical valve replacement: 15 patients undergoing surgical valve replacement (SAVR)
  Interventions: Other: Blood sample
- Patients with aortic stenosis, undergoing transcatheter aortic valve implantation: 15 patients undergoing transcatheter aortic valve replacement (TAVR)
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — After blood sampling, patients will undergo a Color Doppler Echocardiogram, a non-invasive method
  Other Names: Color Doppler echocardiogram

SUMMARY:
The aim of our study is to investigate the effects of impaired left ventricular remodeling on the short- and long-term prognosis in AS partecipants undergoing extracorporeal circulation during valve repair surgery and in partecipants undergoing implantation transcatheter. For the achievement of these purposes, markers obtained from will be considered cardiovascular imaging methods, such as color Doppler echocardiography and isolated biomarkers from peripheral blood and heart tissue.

DETAILED DESCRIPTION:
Participation in this study includes, following enrollment, a visit of follow up (6/12 months) on the occasion of a concomitant medical check-up scheduled according to normal clinical practice. During these visits venous and contextual blood samples will be taken echocardiographic examination for re-evaluation of ejection fraction, as per normal practice clinic. The only variant will be the withdrawal of an additional aliquot of blood during the sampling standard blood.

All enrolled partecipants will undergo the optimal medical treatment provided by current and more recent guidelines for the treatment of heart valve disease. Joining this study will not result any modification of the current therapy, which will be established by the attending physician according to the correct one clinical practice.

ELIGIBILITY:
Inclusion Criteria:

-30 patients with a diagnosis of severe aortic stenosis and preserved ejection fraction to echocardiographic evaluation

Exclusion Criteria:

* inflammatory;
* infectious diseases;
* neoplasms;
* ailments immunological or haematological;
* treatment with anti-inflammatory drugs except aspirin a low dose (75-160 mg);
* age > 85 years;
* advanced chronic kidney disease with filtrate glomerular heart rate (eGFR) estimated by MDRD equation <30 ml/min./1.73 m2.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 patients admitted to our Department will be enrolled in our study of Cardiovascular Sciences with a diagnosis of severe aortic stenosis and preserved ejection fraction echocardiographic evaluation, divided into two categories:
  1. 15 patients undergoing surgical valve replacement (SAVR)
  2. 15 patients undergoing transcatheter aortic valve replacement (TAVR)
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2023-12-13 (Estimated)

PRIMARY OUTCOMES:
Description of the two serum biomarkers of mitochondrial dysfunction | 1 year
  Description of the two serum biomarkers of mitochondrial dysfunction Myeloperoxidase (MPO) and Lactoferrin (LF) and the indices of myocardial performance, systolic and diastolic function of the left ventricle in patients undergoing invasive (SAVR) or non-invasive (TAVR) monitoring.

SECONDARY OUTCOMES:
Evaluation of the correlation between the two serum biomarkers of mitochondrial dysfunction | 6 months
  The two serum biomarkers and the myocardial performance indices, of the left ventricular systolic and diastolic function , evaluated in patients undergoing invasive (SAVR) or non-invasive monitoring (TAVR).
Evaluation of gene expression of molecular pathways involved in ventricular remodeling and correlation with echocardiographic parameters of left ventricular performance. | 6 months
  The gene expression of the molecular pathways involved in ventricular remodeling and the correlation with echocardiographic parameters of left ventricular performance, will be evaluated through methods:
  * peripheral blood sampling
  * immunochemical analysis
  * evaluation of the oxidant and anti-oxidant capacity in vitro

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Gemelli, Roma, Italy

IPD SHARING:
Plan to Share IPD: Yes